CLINICAL TRIAL: NCT03657134
Title: Introductory Clinical Trial for Measuring Patients Before, During, and After an Electrophysiology (EP) Procedure With a Novel, Body-Worn Sensor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-01618
Record Dates: First submitted 2018-08-08; First posted 2018-09-04 (Actual); Results first posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-08

CONDITIONS: Atrial Fibrillation; Ventricular Tachycardia
MeSH Terms: conditions — Atrial Fibrillation; Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- EP Procedure (Experimental): Patient will continuously wear the CoVa-2 monitoring system until they are discharged. During this period, data from the sensor will be sent to the Gateway and Cloud-based System, and then analyzed retrospectively.
  Interventions: Diagnostic Test: CoVa-2 Monitoring System

INTERVENTIONS:
Diagnostic Test: CoVa-2 Monitoring System — Upon completion of EP procedure, CoVa-2 monitoring system will be applied until discharge. Data from the sensor will be sent to the Gateway and Cloud-based system and analyzed retrospectively.

SUMMARY:
Subjects will be consented to wear the CoVa-2 monitoring system prior to (baseline), during, and after an Electrophysiology Procedure (EP). During this time, the system will measure the following parameters from subjects: heart rate (HR), Heart Rate Variability (HRV), respiration rate (RR), and Cardiac Output (CO). Data will be retrospectively analyzed to determine if the system effectively operates under these conditions, and can effectively monitor subjects and allow them to be discharged early from the hospital. Subjects will not be measured while transferred in and out of the operating room. Approximate sample size is 20 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with arrhythmias and other cardiac conditions that are scheduled for EP procedures.
2. Subject is over 22 years of age at the time of consenting
3. Subject and/or legally authorized representative is willing to undergo the informed consent process prior to enrollment in the study

Exclusion Criteria:

1. Pregnant subjects
2. Subjects who are participating in another clinical study that may affect the results of either study
3. Subjects who are unwilling or unable to wear the sensor (and electrodes) for a period of up to 14 hours
4. Subjects who are considered by the principle investigator to be medically unsuitable for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2020-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lior Jankelson, MD, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- EP Procedure: Patient will continuously wear the CoVa TM 2 system until they are discharged for period of about 24 hours. During this period, data from the sensor will be sent to the Gateway and Cloud- based System, and then analyzed retrospectively.
  CoVa 2 Sensor: Upon completion of EP procedure, CoVa 2 sensor will be applied until discharge. Data from the sensor will be sent to the Gateway and Cloudbased system and analyzed retrospectively.
Period: Overall Study
Arm/Group | EP Procedure
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | EP Procedure
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 57 [49 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Average Change in Heart Rate (HR)
Description: HR data is retrospectively analyzed from the CoVa-2 monitoring system, and the average change in HR (prior to the start of EP (baseline) to completion of EP (8 hours)) is reported.
Time Frame: Baseline, 8 Hours
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Groups:
- EP Procedure: Patient will continuously wear the CoVa-2 system until they are discharged for period of about 24 hours. During this period, data from the sensor will be sent to the Gateway and Cloud-based System, and then analyzed retrospectively.
  CoVa-2 Sensor: Upon completion of EP procedure, CoVa 2-sensor will be applied until discharge.
Arm/Group | EP Procedure
Number analyzed (Participants) | 20
beats per minute (bpm) | 6.5 (0.3)

2. Primary Outcome: Average Change in Respiratory Rate (RR)
Description: RR data is retrospectively analyzed from the CoVa-2 monitoring system, and the average change in RR (prior to the start of EP (baseline) to completion of EP (8 hours)) is reported.
Time Frame: Baseline, 8 Hours
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | EP Procedure
Number analyzed (Participants) | 20
bpm | 3.8 (0.8)

ADVERSE EVENTS:
Time Frame: 1 Week
Arm/Group | EP Procedure
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2018-02-20): https://cdn.clinicaltrials.gov/large-docs/34/NCT03657134/Prot_001.pdf